CLINICAL TRIAL: NCT07238816
Title: A Single-centre, Open-label, Randomised, Single-dose Study to Evaluate the Effect of Pre- and Post-dose Meal Timings on the Pharmacokinetic Properties of Inno8 in Healthy Participants
Brief Title: A Research Study Looking at How Food Intake Affects Inno8 in the Body of Healthy People
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7442-8255; Universal Trial Number (Other: U1111-1315-2873)
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Participants will receive oral dose of NNC0442-0344 A.
  Interventions: Drug: NNC0442-0344 A
- Group B (Experimental): Participants will receive oral dose of NNC0442-0344 A.
  Interventions: Drug: NNC0442-0344 A
- Group C (Experimental): Participants will receive oral dose of NNC0442-0344 A.
  Interventions: Drug: NNC0442-0344 A
- Reference dose (Active Comparator): Participants will receive oral dose of NNC0442-0344 A.
  Interventions: Drug: NNC0442-0344 A

INTERVENTIONS:
Drug: NNC0442-0344 A — NNC0442-0344 A will be administered orally.
  Other Names: Inno8

SUMMARY:
The purpose of this study is to test a new medicine called Inno8. The study will test how eating and drinking before and after taking Inno8 affects how well it is absorbed in the stomach. The study consists of four arms. Participants will take the study medicine after an overnight fast. How long participants will need to fast depends on which group participants are in. After taking the study medicine, participants will need to fast again. The study will last for up to 9.5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Age 18-45 years (both inclusive) at the time of signing informed consent.
* Body mass index between 18.5 and 29.9 kilogram per square meter (kg/m^2) (both inclusive) at screening.
* Body weight between 60.0 and 100.0 kilogram (kg) (both inclusive) at screening.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Factor VIII activity greater than or equal to (≥) 150 percentage (%) at screening.
* Increased risk of thrombosis, e.g. known history of personal or first-degree relative(s) with unprovoked deep vein thrombosis.
* Any clinical signs or established diagnosis of venous or arterial thromboembolic disease.
* Any of the thrombophilia markers listed below:
* Lupus anticoagulant, anti-cardiolipin antibody Immunoglobulin G (IgG) and Immunoglobulin M (IgM) or anti-β2 glycoprotein I antibody (IgG and IgM) outside the normal laboratory range at screening.
* Heterozygosity or homozygosity for the factor V Leiden mutation (G1691A) OR heterozygosity or homozygosity for the prothrombin mutation (G20210A) OR compound heterozygosity for the factor V Leiden (G1691A) and prothrombin mutation (G20210A).
* Protein C, protein S or antithrombin below the lower normal laboratory range.
* Any known coagulation disorders.
* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
AUC0-∞: the area under the plasma Inno8 concentration-time curve from time 0 to infinity after a single oral dose | From baseline (Day 1) to day 17
  Measured as nanograms*day per millilitre (ng*day/mL).

SECONDARY OUTCOMES:
Cmax: Maximum observed plasma Inno8 concentration after a single oral dose | From baseline (Day 1) to day 17
  Measured as nanograms per millilitre (ng/mL).
Tmax: The time to maximum observed plasma Inno8 concentration after a single oral dose | From baseline (Day 1) to day 17
  Measured as hours.
Number of treatment emergent adverse events | From time of dosing (Day 1) to day 36
  Measured as count of events.
Change in D-dimer | From baseline (Day 1) to day 36
  Measured as absolute (ng/mL) and percentage (%).
Change in prothrombin fragment 1 and 2 | From baseline (Day 1) to day 36
  Measured as absolute [(picomoles per litre) pmol/L] and %.
Change in fibrinogen | From baseline (Day 1) to day 36
  Measured as absolute [(milligrams per decilitre) mg/dL] and %.
Change in platelets | From baseline (Day 1) to day 36
  Measured as absolute [(ten to the ninth power per litre) 10^9/L] and %.
Change in FIX antigen | From baseline (Day 1) to day 36
  Measured as %.
Change in FX antigen | From baseline (Day 1) to day 36
  Measured as %.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Altasciences Clinical LA, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com